CLINICAL TRIAL: NCT04965051
Title: A Prospective, Randomized, Open-label, Parallel Group Study to Evaluate Safety and Efficacy of Insulin Degludec/Insulin Aspart in Patients With Type 1 Diabetes Mellitus
Brief Title: Safety and Efficacy of Insulin Degludec/Insulin Aspart in Patients With T1DM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0407
Record Dates: First submitted 2021-07-07; First posted 2021-07-16 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: Type 1 Diabetes Mellitus With Diabetic Gastroparesis; HbA1c; Time in Range
Keywords: Type 1 Diabetes; insulin degludec/insulin aspart; HbA1c; Time in Range
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — insulin degludec; Insulin Aspart; insulin degludec, insulin aspart drug combination; Insulin Detemir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IDegAsp group (Experimental): IDegAsp twice daily
  Interventions: Drug: insulin degludec/insulin aspart (IDegAsp)
- basal insulin plus pre-prandial insulin group (Active Comparator): basal insulin once or twice daily plus pre-prandial insulin
  Interventions: Drug: basal insulin plus pre-prandial insulin

INTERVENTIONS:
Drug: insulin degludec/insulin aspart (IDegAsp) — To evaluate the efficacy and safety of the IDegAsp in T1DM
  Other Names: Ryzodeg
  Arms: IDegAsp group
Drug: basal insulin plus pre-prandial insulin — To evaluate the efficacy and safety of basal insulin plus pre-prandial insulin in T1DM
  Other Names: Levemir/Lantus/Tresiba plus NovoLog/Humalog/Apidra
  Arms: basal insulin plus pre-prandial insulin group

SUMMARY:
In this prospective, randomized, open-label, parallel group trial, the safety and efficacy of insulin degludec/insulin aspart (IDegAsp) twice daily will be compared with basal insulin once or twice daily plus pre-prandial insulin after 16 weeks of treatment in patients with type 1 diabetes. This trial will enable assessment of the clinically relevant endpoint of a change in HbA1c and Time in Range (TIR).

DETAILED DESCRIPTION:
The objective of the current study is to investigate the efficacy and safety of IDegAsp twice daily compared to basal insulin once or twice daily plus pre-prandial insulin for 16 weeks in patients with type 1 diabetes mellitus. The primary endpoint in this study is the change from baseline in HbA1c. Patients with type 1 diabetes who meet the entry criteria are planned for inclusion in this trial. Approximately 40 patients will be enrolled in the study. Patients who qualify will be randomized to IDegAsp group or basal plus pre-prandial insulin group. Duration of treatment includes 2-week screening period, 16-week treatment observation period and 1-week follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 and ≤75 years with type 1 diabetes;
* Diagnosed as T1DM ≥ 12 months before enrollment in the study;
* HbA1c ≥ 7.0 to ≤10.0%;
* Receipt of basal plus pre-prandial insulin and/or oral anti-diabetic agents ≥ 12 weeks before enrollment in the study;
* BMI ≤ 35kg / m2.

Exclusion Criteria:

* Patients with any of the following conditions will be excluded:
* Pregnant or lactating women
* Severe hypoglycemia within one month;
* Myocardial infarction, stroke or other severe cardiovascular events within 6 months prior to informed consent
* Receipt of Sulfonylureas, Meglitinides derivatives, Thiazolidinediones, Dpp-4 inhibitors or GLP-1 agonists within 3 months prior to informed consent;
* Current treatment with systemic steroids or immunosuppressive agents, or have immunologic deficiency disease at time of informed consent
* Severe mental instability, or alcohol abuse, or drug abuse
* Cancer within 5 years prior to informed consent
* Pancreatitis of severe infectious diseases within 1 months prior to informed consent
* Known hypersensitivity or allergy to the insulin
* Renal impairment (CKD-EPI eGFR<60ml/min)
* Impaired hepatic function, defined by serum levels of either ALT (SGPT), AST (SGOT), or alkaline phosphatase above 3 x upper limit of normal (ULN) as determined
* Participation in another trial within 2 months prior to informed consent
* Patients that investigators believe may fail to complete the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-08 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
HbA1c | 16 weeks
  the change from baseline in HbA1c after 16 weeks of treatment in all patients

SECONDARY OUTCOMES:
Time In Range (TIR) | 16 weeks
  The change from baseline in Time in Range (3.9-10mmol/L) after 16 weeks of treatment in all patients (using flash continuous glucose monitoring (FCGM)).
Time to occurrence of treat to target | 16 weeks
  Fasting glucose on treatment <7mmol/L and non-fasting glucose <10mmol/L, or TIR >70%) (SMBG or FCGM)
Occurrence of a treat to target response and without any hypoglycemic episodes | 16 weeks
  Occurrence of a treat to target response and without any hypoglycemic episodes
EQ-5D Health Questionnaire | 16 weeks
  the EQ-5D descriptive system The change from baseline after 16 weeks of treatment
Short Form 36 (SF-36) | 16 weeks
  The change from baseline after 16 weeks of treatment
Insulin dose | 16 weeks
  The change from baseline after 16 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Yuezhong Ren, MD, Principal Investigator — 2nd Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No